CLINICAL TRIAL: NCT02047578
Title: Targeted Busulfan, Fludarabine, Etoposide Conditioning Regimen for Hematopoietic Stem Cell Transplantation in Childhood and Adolescent Acute Lymphoblastic Leukemia
Brief Title: Targeted Busulfan, Fludarabine, Etoposide Conditioning Regimen for HSCT in Childhood and Adolescent ALL.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUCH_ALL_BuFluVP
Record Dates: First submitted 2014-01-09; First posted 2014-01-28 (Estimated); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: hematopoietic stem cell transplantation
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Busulfan (Experimental): Drug: Busulfan First dose: busulfan (120 mg/m2 ivs once daily) (if age<1 yr: 80 mg/ m2) Second to forth dose: according to the daily pharmacokinetic study
  Interventions: Drug: Busulfan

INTERVENTIONS:
Drug: Busulfan — First dose: busulfan (120 mg/m2 ivs once daily) (if age<1 yr: 80 mg/ m2) Second to forth dose: according to the daily pharmacokinetic study

SUMMARY:
To evaluate the outcome of hematopoietic stem cell transplantation using targeted busulfan, fludarabine, etoposide conditioning regimen in childhood and adolescent ALL.

DETAILED DESCRIPTION:
Busulfan is a highly toxic drug with narrow therapeutic window used for the conditioning of hematopoietic stem cell transplantation. High exposure is associated with systemic toxicity such as veno-occlusive disease (VOD) and underexposure is associated with graft failure or relapse. In this study the investigators plan to improve the outcome of hematopoietic stem cell transplantation by using optimal busulfan dose through pharmacokinetic study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are diagnosed as ALL.
2. Patients who need hematopoietic stem cell transplantation
3. Age: up to 21 years
4. Performance status: ECOG 0-2.
5. Patients must be free of significant functional deficits in major organs, but the following eligibility criteria may be modified in individual cases. 1. Heart: a shortening fraction > 30% and ejection fraction > 45%. 2. Liver: total bilirubin < 2 × upper limit of normal; ALT < 3 × upper limit of normal. 3. Kidney: creatinine <2 × normal or a creatinine clearance (GFR) > 60 ml/min/1.73m2.
6. Patients must lack any active viral infections or active fungal infection.
7. Appropriate donor is available: Matched in 6/6 of A, B, DR loci.
8. Patients (or one of parents if patients age < 19) should sign informed consent.

Exclusion Criteria:

1. Pregnant or nursing women.
2. Malignant or nonmalignant illness that is uncontrolled or whose control may be jeopardized by complications of study therapy.
3. Psychiatric disorder that would preclude compliance.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Estimated)
Dates: Start 2014-02-05 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
1-year event free survival after hematopoietic stem cell transplantation. | at 1 year
  To evaluate 1-year event free survival after hematopoietic stem cell transplantation.

SECONDARY OUTCOMES:
Engraftment rate | 1, 3, 6 and 12 months after transplantation
  To evaluate engraftment rate

OTHER OUTCOMES:
Toxicities associated with hematopoietic stem cell transplantation | 1, 3, 6 and 12 months after transplantation
  To evaluate toxicities associated with hematopoietic stem cell transplantation. Toxicities will be assessed with number of participants.
Acute GVHD | 1, 3, 6 and 12 months after transplantation
  To evaluate acute GVHD
Chronic GVHD | 1, 3, 6 and 12 months after transplantation
  To evaluate chronic GVHD
Treatment related mortality | 1, 3, 6 and 12 months after transplantation
  To evaluate treatment related mortality
Relapse rate | 1, 3, 6 and 12 months after transplantation
  To evaluate relapse rate

CONTACTS AND LOCATIONS:
Overall Officials: Hyoung Jin Kang, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Daehangno, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided